CLINICAL TRIAL: NCT04160858
Title: Effects of the Spinal Cord Injury Exercise Guidelines on Pain: A Randomized Controlled Trial
Brief Title: Effects of Spinal Cord Injury Exercise Guidelines
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kathleen Martin Ginis, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCI Ex Guidelines Pain: RCT
Record Dates: First submitted 2019-08-16; First posted 2019-11-13 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Chronic Pain; Spinal Cord Injuries
MeSH Terms: conditions — Chronic Pain; Spinal Cord Injuries | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The trial design is a two-arm, single-blinded ( i.e. assessors and analysts blinded to allocation), RCT with a 6-month intervention period and 6-month follow-up (Exercise condition only). After baseline assessments, participants will be randomly allocated to 6 mos of exercise ("Exercise") or a wait-list ("Control") using a 1:1 ratio. The trial is designed to be comparable to usual care and maximize PRECIS scores, while providing insight on mechanisms that may explain intervention effects.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Keeping outcome assessors and data analysts blinded to the allocation (i.e. participants and groups identifiable by number only). This ensures unbiased ascertainment and analysis of outcomes. When participants arrive at the lab for testing, they will be instructed not to reveal their allocated condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Condition (Experimental): The intervention is a personalized exercise prescription based on the International Scientific Spinal Cord Injury (SCI) Exercise Guidelines. Participants begin at the Starting Level guideline: 20 min aerobic exercise, 2x/wk, at 70% of heart rate reserve (or a Borg Continuous Ratio 0-10 rating of 6), & 3 sets of 10 repetitions of strengthening exercises (each major functioning muscle group at 50-80% of 1-rep max), 2x/wk. Participants will gradually increase aerobic exercise to 30 min, 3x/wk (i.e. the Advanced Level guideline). Exercise implementation will be supported by a fitness trainer and an exercise counsellor with SCI-specific training and experience.
  Interventions: Other: Exercise
- Wait-list Control (Active Comparator): Control participants will not get an exercise prescription. They will be asked to refrain from lifestyle changes for 6 mos. After the 6-month waitlist period, Controls will receive the same resources as Exercisers.
  Interventions: Other: Control

INTERVENTIONS:
Other: Exercise — Spinal Cord Injury Exercise Guidelines: Participants will begin at the Starting Level which is 20 mins of moderate to vigorous aerobic activity 2x/week & 3 sets of 10 repeats of strength training 2x/week. They will progress to Advanced Level which is 30 mins of moderate to vigorous aerobic activity 3x/week and 3 sets of 10 repetitions of strength training 2x/week. The intervention duration is 6 months.
  Arms: Exercise Condition
Other: Control — Wait-list control
  Arms: Wait-list Control

SUMMARY:
Over 85,000 Canadians live with a spinal cord injury (SCI). The vast majority experience chronic pain from neuropathic or musculoskeletal origins, with many reporting the pain to be more physically, psychologically and socially debilitating than the injury itself. Currently, pharmaceuticals are the front line treatment recommendation for SCI pain, despite having many side-effects and giving minimal relief. Alternatively, studies conducted in controlled lab and clinical settings suggest that exercise may be a safe, effective behavioural strategy for reducing SCI-related chronic pain. Two ways in which exercise may alleviate pain are by reducing inflammation and increasing descending inhibitory control. To date, no study has tested the effects of exercise, performed in a home-/community-setting, on chronic pain in adults with SCI. Furthermore, information on the exercise dose required to alleviate chronic SCI pain is virtually non-existent, making it impossible for clinicians and fitness trainers to make evidence- informed recommendations regarding the types and amounts of exercise to perform in order to manage SCI pain. Recently (2018), an international team published two scientific SCI exercise guidelines: one to improve fitness and one to improve cardiometabolic health. These scientific guidelines have been translated into Canadian community SCI exercise guidelines and provide the exercise prescription for the proposed study.

The investigators' overarching research question is: can home-/community-based exercise-prescribed according to these new SCI exercise guidelines and supported through a theory-based behavioural intervention- significantly reduce chronic pain in adults with SCI?

DETAILED DESCRIPTION:
PROPOSED TRIAL. Using an integrated knowledge translation framework (iKT), the primary aim of this pragmatic Randomized Controlled Trial (RCT) is to examine the effects of 6 months of home-/community-based exercise, prescribed according to the SCI exercise guidelines, on chronic bodily pain experienced by adults with SCI. Secondary aims are to test for 1) differential effects on musculoskeletal and neuropathic pain; 2) changes in inflammation and inhibitory control as pathways by which exercise reduces pain; 3) effects of chronic pain reductions on subjective well-being; and 4) economic benefits of the intervention.

TRIAL MANAGEMENT. The experienced team of researchers has SCI-specific expertise in exercise psychology and physiology, pain and physiatry as well as health sciences expertise in immunology, biostatistics, health economics, and pragmatic RCT design and management. The team includes knowledge users representing local, provincial and national organizations, and a collaborator with lived experience of SCI.

SIGNIFICANCE. The investigators' novel idea is that home-/community-based exercise performed according to the SCI exercise guidelines can be an effective behavioural strategy for reducing chronic pain in adults with SCI. Critically, this will be the first SCI exercise RCT to use chronic bodily pain as the primary outcome and to assess potential pathways by which exercise may alleviate pain. Furthermore, this will be the first pragmatic RCT of exercise as a behavioural pain management strategy conducted among adults with SCI. Importantly, our community-engaged, iKT approach will ensure rapid translation and dissemination of findings to Canadian and international end-users including clinicians, fitness programmers, people living with SCI and the community organizations that support them.

ELIGIBILITY:
Inclusion Criteria:

* (i) adults aged >18 with an spinal cord injury (SCI), traumatic or non-traumatic cause;
* (ii) ASIA impairment scale classifications A-D, injury levels C3 or below;
* (iii) >12 mos post-injury [criteria i-iii capture the group to whom the SCI Exercise Guidelines apply);
* (iv) reporting chronic pain, defined as pain that persists or recurs for more than 3 mos on a question taken from the US Model SCI Systems measures: ["Using a 0 to 10 scale with 10 being pain so severe you could not stand it and 0 being no pain, what has been the usual level of pain over the past 3 months?"] and scoring at or above 1;
* (v) report pain secondary to SCI that is classified as neuropathic and/or musculoskeletal (MSK) using theInternational SCI Pain Basic Data Set (v2.0) pain descriptions. [The trial physiatrist will train the research coordinators to use the Data Set and will make final decisions on unclear cases.];
* (vi) report <40 min/wk of structured, moderate intensity, aerobic exercise and <2 bouts/week of strength training (i.e. less than the Starting Level guideline) on a modified version of the Leisure Time Physical Activity Questionnaire-SCI (<15% of Canadians with SCI currently achieve the Starting Level so the trial can assess the effects of increasing exercise to recommended levels;
* (vii) no medical contra-indications to performing a maximal exercise test;
* (viii) have access to a phone.

Exclusion Criteria:

* (i) chronic pain with exclusively non-MSK or non-neuropathic origins (e.g. headache, abdominal pain-because the effects of exercise on these pain types are unknown);
* (ii) insufficient diaphragmatic control and arm functioning to do upper-body exercise;
* (iii) live beyond driving distance of the research site;
* (iv) insufficient English language proficiency to complete questionnaires and converse with the fitness trainer and counselor;
* (v) have been previously told s/he has a cognitive or memory impairment;
* (vi) pregnant (because safety of the guidelines are unknown);
* (vii) hospital in-patient at the time of enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2025-02-14 (Estimated); Study Completion 2025-02-14 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline, between and within group comparison, in Bodily Pain | Baseline, 3 months, 6 months
  Outcome Measure - SF-36 Bodily Pain (SF-36 Pain) subscale to assess pain severity and interference. Lower scores indicated greater bodily pain (0-100 total score range).

SECONDARY OUTCOMES:
International Spinal Cord Injury Pain Basic Data Set v2.0 | Baseline, 3 months, 6 months
  Measures overall interference of musculoskeletal and neuropathic pain, as well as the intensity of each specific pain location and type (up to three pain problems).
Presence of Neuropathic Pain | Baseline, 3 months, 6 months
  Outcome Measure: Neuropathic Pain Diagnostic Questionnaire (DN-4) (total score range 0-10 with scores ≥ 4 indicating neuropathic pain).
Inhibitory Control of Pain assessed by Conditioned Pain Modulation | Baseline, 3 months, 6 months
  This test measures the extent to which the application of a painful conditioning stimulus changes the perceived painfulness of a test stimulus. The test stimulus will be delivered by using a pressure algometer (contact area 1 cm2; Algomed Computerized Algometry; Medoc AMS), whereby the threshold for pressure induced pain will be measured on an upper extremity site that has sensory innervation, in 3 series of slowly increasing stimulus intensities (0.5 kg/s, corresponding to ca. 50 kPa/s). Participants will report the instant when pain is initially perceived, over and above the application of pressure. Pain threshold will be determined as the arithmetic mean of the 3 series (in kPA). Inhibitory control is calculated as the change in pain ratings for the test stimulus, from before to after application of the conditioning stimulus (bigger decreases in pain ratings indicate better inhibitory control/pain modulation).
Fasting plasma concentrations of cytokines IL-6 | Baseline, 3 months, 6 months
  Outcome Measure Blood Sampling - A fasting blood sample (>12 h) will be taken from the antecubital vein. IL-6 will be measured by high-sensitivity ELISA (R&D Quantikine); fasting glucose (ADVIA1650, Siemens) and insulin (Roche Diagnostics, Mannheim, Germany) by automated clinical analyzers to calculate the corresponding homeostatic model assessment index; and triglycerides, total cholesterol and HDL cholesterol using an ADVIA 1650 chemistry system, after which LDL cholesterol is calculated.
Fasting plasma concentrations of cytokines TNF-α | Baseline, 3 months, 6 months
  Outcome Measure Blood Sampling- A fasting blood sample (>12 h) will be taken from the antecubital vein. TNF-α will be measured by high-sensitivity ELISA (R&D Quantikine); fasting glucose (ADVIA1650, Siemens) and insulin (Roche Diagnostics, Mannheim, Germany) by automated clinical analyzers to calculate the corresponding homeostatic model assessment index; and triglycerides, total cholesterol and HDL cholesterol using an ADVIA 1650 chemistry system, after which LDL cholesterol is calculated.
Subjective Well-being: Perceived Stress | Baseline, 3 months, 6 months
  Outcome Measure - Perceived Stress Scale. Lower scores indicated lower perceived stress (0-40 total score range)
Subjective Well-being: Quality of Life | Baseline, 3 months, 6 months
  Outcome Measure - SCI-QOL (Quality of Life) measurement system which measures of Positive Affect and Well-Being (scale range 10-50; higher scores greater positive affect and wellbeing), and Satisfaction with Social Roles and Activities (scale range 10-50; higher scores indicate greater satisfaction in social roles and activities) .
Subjective Well-being: Life Satisfaction | Baseline, 3 months, 6 months
  Outcome Measure - Diener's Satisfaction with Life Scale. Scale range 5-35 with higher scores indicating greater life satisfaction.
Subjective Well-being: Experiential Aspects of Participation | Baseline, 3 months, 6 months
  Outcome Measure: Measure of Experiential Aspects of Participation (MeEAP). This questionnaire measures Autonomy, Belongingness, Challenge, Engagement, Mastery and Meaning as experiential aspects of participation (score ranges 1-7 with higher scores indicating better participation experiences).
Economic Evaluation: Health Care Costs | Baseline, 3 months, 6 months
  Outcome Measure - Health Care Utilization questionnaire (7 questions asking if and who they received health care care from, why and why not) Reference: Luc Noreau, Vanessa K. Noonan, John Cobb, Jean Leblond, Frédéric S. Dumont. Spinal Cord Injury Community Survey: A National, Comprehensive Study to Portray the Lives of Canadians with Spinal Cord Injury. Top Spinal Cord Inj Rehabil. 2014 Fall; 20(4): 249-264. Published online 2014 Oct 30. doi: 10.1310/sci2004-249
Health-related Quality of Life | Baseline, 3 months, 6 months
  Outcome Measure - 5 level version of EuroQol-5D (EQ-5D). Overall scale range 5-25 with a lower score indicating a higher quality of life.
Capability Wellbeing | Baseline, 3 months, 6 months
  Outcome Measure - an Index of Capability for Adults (ICECAP-A). Overall scale range 5-20 with a lower score indicating a lower index of capability in life.
Inflammation Fidelity Checks | Baseline, 3 months, 6 months
  Check/control for acute infection that may influence inflammatory markers in the sample, a complete blood count will be performed.
Intervention Fidelity Check: Peak power output over max aerobic arm crank test | Baseline, 3 months, 6 months
  Outcome Measure - progressive arm crank test to exhaustion using a Lode arm crank ergometer (Groningen, the Netherlands) and metabolic cart (TrueOne® 2400, ParvoMedics,Utah) [average max 30-s Watts produced, i.e. >0 W)
Intervention Fidelity Check: 1 Repetition-Maximum strength test bench press | Baseline, 3 months, 6 months
  Outcome Measure - Multiple trials of 1-rep max bench press tests (to minimise learning effects as per the latest strength measurement guidelines) using HUR strength equipment (Kokkola, Finland) - [max Force produced, measured in kg, i.e. >0 W)
Intervention Fidelity Check : Peak oxygen uptake over max aerobic arm crank test | Baseline, 3 months, 6 months
  Outcome Measure - progressive arm crank test to exhaustion using a Lode arm crank ergometer (Groningen, the Netherlands) and metabolic cart (TrueOne® 2400, ParvoMedics,Utah) - [average 30-s peak oxygen uptake measured, i.e. >0 L/min and >0 L/min/kg body mass)
Intervention Fidelity Check : 1 Repetition-Maximum strength test seated row | Baseline, 3 months, 6 months
  Outcome Measure - and multiple trials of 1-rep max seated row tests (to minimise learning effects as per the latest strength measurement guidelines) using HUR strength equipment (Kokkola, Finland) - [max Force produced, measured in kg, i.e. >0 W)

OTHER OUTCOMES:
Fidelity of the fitness trainer and exercise counselor to their protocols | Weekly during the intervention for the exercise group (24 weeks)
  To assess fidelity of the fitness trainer and exercise counselor to their protocols, similar to our previous studies, both will complete checklists during each session which will be reviewed by the NPA. The NPA will also make random checks of a subset of audio recordings of counseling sessions and real-time visits to the fitness training sessions. If deviations from the protocol occur, the NPA will provide corrective feedback.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Martin Ginis, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No